CLINICAL TRIAL: NCT06091553
Title: Comparison of the Efficacy and Safety of Duloxetine Augmented With Gabapentin and Duloxetine Augmented With Amitriptyline vs Duloxetine Alone in Chemotherapy -Induced Neuropathy: A Randomized Controlled Trial
Brief Title: Comparison of the Efficacy and Safety of Duloxetine Augmented With Gabapentin and Duloxetine Augmented With Amitriptyline vs Duloxetine Alone in Chemotherapy -Induced Neuropathy
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Beni-Suef University (Other)
Responsible Party: Principal Investigator, Hager salah el din, Principal Investigator, Beni-Suef University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IORG0006240
Record Dates: First submitted 2023-10-14; First posted 2023-10-19 (Actual); Last update posted 2024-04-16 (Actual); Status verified 2024-04

CONDITIONS: Neuropathy in Cacer Patien
MeSH Terms: interventions — Duloxetine Hydrochloride; Gabapentin; Amitriptyline

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Duloxetine alone (as monotherapy) (Active Comparator): Duloxetine alone (as monotherapy)
  Interventions: Drug: Duloxetine alone
- Duloxetine augmented with gabapentin (as combined therapy) (Active Comparator): Duloxetine augmented with gabapentin (as combined therapy)
  Interventions: Drug: Duloxetine augmented with gabapentin
- Duloxetine augmented with amitriptyline (as combined therapy) (Active Comparator): Duloxetine augmented with amitriptyline (as combined therapy)
  Interventions: Drug: Duloxetine augmented with amitriptyline (as combined therapy)
- control (No Intervention): control

INTERVENTIONS:
Drug: Duloxetine alone — 30 mg once daily for 1 week, then 60 mg once daily
  Arms: Duloxetine alone (as monotherapy)
Drug: Duloxetine augmented with gabapentin — 30 mg once daily for 1 week, then 60 mg once daily 300 mg at bedtime
  Arms: Duloxetine augmented with gabapentin (as combined therapy)
Drug: Duloxetine augmented with amitriptyline (as combined therapy) — 10 to 25 mg once daily at bedtime 30 mg once daily for 1 week, then 60 mg once daily
  Arms: Duloxetine augmented with amitriptyline (as combined therapy)

SUMMARY:
This study aimed to elucidate the relationship between the Efficacy and Safety of Comparison of the Efficacy and Safety Duloxetine augmented with gabapentin and amitriptyline augmented with Duloxetine vs duloxetine alone in chemotherapy -Induced Neuropathy in cancer patients.

ELIGIBILITY:
Inclusion Criteria:

* -Patients of any age must have histologically or cytologically confirmed cancer by the Laboratory of Pathology.
* Patients must sign an informed consent form (ICF) voluntarily and be able to understand and comply with the requirements of the study;
* Patients must be 18 to 75 years of age (including cut-offs) on the date of signing the informed consent form, regardless of gender;
* Patients must received treatment with a chemotherapy regimen .
* Patients must have ≥ grade 1 sensory chemotherapy-induced peripheral neuropathy (CIPN) with NRS ≥ 4/10 according to the NCI Common Toxicity Criteria for Adverse Events (CTCAE) v.5.0 grading scale
* Eastern Cooperative Oncology Group performance status (ECOG PS): 0-2;
* Expected survival of ≥ 3 months
* There is no maximum number of prior medical therapies.

Exclusion Criteria:

* History of allergic reactions attributed to compounds of similar chemical or biologic composition to duloxetine, amitriptyline and gabapentin
* Pregnant women are excluded from this study.
* Life expectancy less than 6 months
* Inability or unwillingness to comply with research protocols.
* Patients with the presence of active brain or meningeal metastases.
* Patients with the presence of uncontrolled closed-angle glaucoma.
* Patients with the presence of neuropathy caused by any type of nerve compression as diabetes.
* The presence of mental illness, epilepsy, mania, suicidal depression, dementia or alcohol or drug abuse that may have an impact on compliance with trial requirements.
* The presence of comorbid cardiovascular disease, including but not limited to: (1) New York Heart Association (NYHA) criteria ≥ grade 2 heart failure; (2) severe/unstable angina pectoris; (3) myocardial infarction or cerebrovascular accident within 6 months prior to first dose; (4) atrial fibrillation and supraventricular or ventricular arrhythmias requiring treatment; (5) pre-existing symptomatic superior vena cava syndrome; (6) corrected QT interval (QTc) > 450 ms (men); QTc > 470 ms (women); (7) hypertensive disease not controlled by antihypertensive medication: systolic blood pressure ≥ 140 mmHg or diastolic blood pressure ≥ 90 mmHg;
* Patients with other medical history or evidence of disease that has the potential to confound trial results are excluded from the study,

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2023-10-10 (Actual); Primary Completion 2024-09-30 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
The difference in numerical rating scale (NRS) daily pain measured during the final follow-up week (week 8) between the treatments. | 8 week

SECONDARY OUTCOMES:
Quality of Life Score | 8 week
Anxiety and depression Score | 8 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Beni-Seuf University Hospital, Banī Suwayf, Egypt

IPD SHARING:
Plan to Share IPD: Undecided